CLINICAL TRIAL: NCT02190786
Title: Phase II Exploratory Clinical Study of KUX-1151
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KUX1201
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Hyperuricemia
Keywords: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

ARMS (3):
- KUX-1151, Low dose (Experimental)
  Interventions: Drug: KUX-1151
- KUX-1151, Middle dose (Experimental)
  Interventions: Drug: KUX-1151
- KUX-1151, High dose (Experimental)
  Interventions: Drug: KUX-1151

INTERVENTIONS:
Drug: KUX-1151

SUMMARY:
The purpose of this study is to investigate the efficacy, safety and pharmacokinetics of multiple oral administration of KUX-1151 in patients with hyperuricemia including gout.

ELIGIBILITY:
Inclusion Criteria:

* Japanese HU patients (Outpatient)
* Patients who meet the following criteria concerning serum uric acid levels at the screening [1) Gout: > 7.0 mg/dL, 2) HU with complications: ≥ 8.0 mg/dL, 3) HU without complications: ≥ 9.0 mg/dL]

Exclusion Criteria:

* Patients who have any symptom of gouty arthritis within 2 weeks of investigational product administration

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving serum uric acid level ≤ 6 mg/dL | 14 weeks
Percent change from baseline in serum uric acid level | 14 weeks
Change from baseline in serum uric acid level | 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo and Other Japanese City, Japan